CLINICAL TRIAL: NCT00855543
Title: Phospholipase A2 Producing Bacteria, Age at Gestation, Cervical Length Measurement and the Incidence of Pre-Term Labor
Brief Title: Phospholipase A2 Producing Bacteria and Pre-Term Labor
Status: Completed | Type: Observational
Sponsor: CAMC Health System (Other)
Responsible Party: Dr. Byron C. Calhoun, M.D., Charleston Area Medical Center/West Virginia University
Other Study IDs: 08-11-2097
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to better understand (1) if phospholipase A2 producing microorganisms and cytokines (IL-1, IL-4, IL-6, IL-10, and IL-13) are associated with premature labor (2) if pregnant teens are more likely to have phospholipase A2 producing bacteria than a pregnant adults and (3) if there is a difference in the cytokines between pregnant teens and adults.We hypothesize that phospholipase producing microorganisms may trigger the onset of premature labor. The following are hypothesized: (a) The microorganism cultured should show high activities of phospholipase A2 (b) The cervical length measurement predictive value should correspond to the gestation age at term (c) Vaginal flora of teen will be more susceptible to colonization with higher phospholipase A2 producing bacteria than that of an adult (d) The maternal genotype contribution to the concentration of IL-1, IL-4, IL-6, IL-10, IL-13, and TNF-alpha during the first trimester of pregnancy in teens is different in the production of inflammatory cytokines and modulators(e) The maternal genotype of teens therefore influences the production of phospholipase A2 and causes an increase in preterm delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age <34 weeks
2. Singleton gestation
3. Urinalysis and urine culture collected via clean catch
4. Age range 14 - 45
5. Patient receiving prenatal care at CAMC Women's Medicine Center

Exclusion Criteria:

1. In labor or with uterine contractions
2. Known fetal anomalies
3. Cerclage
4. Dark amniotic fluid suggestive of previous bleeding
5. Multiple gestation
6. Known unbalance chromosomal complement
7. Pregnant patient with prior history of excisional cervical biopsy (either cold knife, loop electrosurgical excision procedure, or laser conization)
8. Patient with mullerian anomaly
9. Patient with 2 or more D&E secondary to spontaneous or induced abortion

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Obstetric patients in West Virginia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byron C Calhoun, MD, Principal Investigator — West Virginia Univeristy/Charleston Area Medical Center
Locations (1):
- Charleston Area Medical Center/West Virginia University, Charleston, West Virginia, United States